CLINICAL TRIAL: NCT04121143
Title: Multicenter, Placebo-controlled, Parallel-randomized, Double-blind, Phase II Study to Investigate the Efficacy, Safety, Tolerability and Pharmacokinetics of SHR-1314 Injection With Moderate to Severe Plaque Psoriasis in Adults
Brief Title: A Clinical Study of SHR-1314 Injection in the Treatment of Moderate to Severe Plaque Psoriasis in Adults
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor's decision
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHR-1314-202
Record Dates: First submitted 2019-09-27; First posted 2019-10-09 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Plaque Psoriasis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Treatment group A (Active Comparator): SHR-1314 low dose short intervals of subcutaneous injection
  Interventions: Biological: IL-17A Antagonist
- Treatment group B (Active Comparator): SHR-1314 high dose long intervals of subcutaneous injection
  Interventions: Biological: IL-17A Antagonist; Biological: Placebos
- Treatment group C (Active Comparator): SHR-1314 high dose short intervals of subcutaneous injection
  Interventions: Biological: IL-17A Antagonist; Biological: Placebos
- Placebo group (Placebo Comparator): Placebo was subcutaneously injected into the 16 weeks turnover SHR-1314 subcutaneous injection
  Interventions: Biological: IL-17A Antagonist; Biological: Placebos

INTERVENTIONS:
Biological: IL-17A Antagonist — SHR-1314 subcutaneous injection
  Other Names: SHR-1314
Biological: Placebos — placebo subcutaneous injection to maintain consistency and to prevent blindness
  Arms: Placebo group; Treatment group B; Treatment group C

SUMMARY:
This is a multicenter, placebo-controlled, parallel-randomized, double-blind, phase II study to investigate the efficacy, safety, tolerability and Pharmacokinetics of SHR-1314 injection with moderate to severe plaque psoriasis in adults

DETAILED DESCRIPTION:
This study was a multicenter, parallel, randomized, double-blind, placebo-controlled clinical trial designed to evaluate the efficacy ,safety, tolerance, and pharmacokinetics (PK) of different SHR-1314 dosing regimens in moderate to severe chronic plaque psoriasis in adults.

ELIGIBILITY:
* Inclusion Criteria:
* Provide written informed consent before any study assessment is performed.
* Male or female at least 18 years of age at screening.
* Chronic plaque psoriasis history ≥ 6 months;At the time of randomization, moderate to severe plaque psoriasis.
* Subject is a candidate for systemic psoriasis therapy and/or phototherapy and/or chemo phototherapy.
* The body mass index (BMI) was ≥18 kg/m2 and ≤35 kg/m2 at screening.
* Exclusion Criteria:
* Diagnosis of psoriasis at screening is not chronic plaque psoriasis
* Severe infection or systemic infection before baseline
* There are other skin problems that researchers believe will hinder the evaluation of psoriasis.
* Subject has a history or symptom of malignancy within 5 years prior to screening, regardless of whether or not treatment has been received, with or without signs of recurrence or metastasis.
* The investigators believe that the subject is not suitable for any clinical condition involved in the clinical study.
* Those who are allergic to the study ingredients or excipients, or who are allergic to other biological agents.
* There is evidence that hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) confirmation test is positive.
* Subject's medical history, symptoms and examination results suggest active tuberculosis or latent tuberculosis.
* Laboratory tests have clinical implications at screening, and the investigators believe that participation in the study may pose unacceptable risks to the subject or impede data analysis.
* Women who are pregnant or breastfeeding at screening or at baseline
* The investigator believes that it will prevent the subject from following and completing any other circumstances of the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-11-09 (Actual); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-30 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects reach to PASI 75 response at 16 weeks | 16 week
  Proportion of subjects with a Psoriatic Area and Severity Index (PASI) score improved by at least 75% (to achieve a PASI 75 response) relative to the baseline PASI score at Week 16

SECONDARY OUTCOMES:
Proportion of subjects achieving PASI 90 response at week 16 | 16 week
  Proportion of subjects with a Psoriatic Area and Severity Index (PASI) score improved by at least 90% (to achieve a PASI 90 response) relative to the baseline PASI score at Week 16 will be evaluated.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Hengrui Pharmaceutical Co., Ltd., Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No